CLINICAL TRIAL: NCT02444520
Title: Persistent Physical Symptoms Reduction Intervention: a Systems Change and Evaluation (PRINCE) - Integrated GP Care for Persistent Physical Symptoms: a Feasibility & Cluster Randomised Controlled Trial
Brief Title: PRINCE Primary: Integrated GP Care for Persistent Physical Symptoms - a Feasibility & Cluster Randomised Controlled Trial
Acronym: PRINCE Primary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: STR130202 (Primary)
Record Dates: First submitted 2015-04-22; First posted 2015-05-14 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2018-08

CONDITIONS: Persistent Physical Symptoms
Keywords: Medically unexplained symptoms; Primary care; Cognitive behaviour therapy skills; Cluster randomised controlled trial; Feasibility
MeSH Terms: conditions — Medically Unexplained Symptoms

STUDY DESIGN:
Intervention Model Description: PRINCE Primary is a cluster randomised waiting list controlled trial to evaluate the acceptability and feasibility of an integrated approach to care in general practice for adults with PPS.
Who Masked: Outcomes Assessor
Masking Description: Patients and GPs will not be blind to treatment allocation due to the nature of the trial (i.e. therapy trial). The trial team member responsible for treatment allocation will be unblind. All outcome data are based on self-report and will be collected either by post or email. The research assistant(s) responsible for contacting participants who have not returned or completed follow-up questionnaires will be unblind. Moreover, the Data Monitoring and Ethics Committee (DMEC), research workers and trial statisticians will remain blind to treatment allocation.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrated GP Care (Experimental): * GP training in utilising cognitive behavioural skills during 10-minute consultations;
  * GP Supervision;
  * Audio-visual and written materials/guidelines for GP's;
  * Copies of self-help materials for patients;• Integrated case management discussion prior to secondary care referral. GPs will be encouraged to consult with a colleague before making a referral;
  * Booklets for patients once consent gained.
  Interventions: Behavioral: Integrated GP Care
- Waiting List Control Group (No Intervention): Patients in the waiting list control group will continue to receive treatment as usual (TAU), and will be crossed over to receive 'Integrated GP Care' at 6 months post randomization.

INTERVENTIONS:
Behavioral: Integrated GP Care — The overall aims of the intervention are to help the patient:
  1. develop an understanding of the relationship between cognitive, emotional, physiological and behavioral aspects of their problem;
  2. understand factors that may be maintaining the problem;
  3. learn how to modify the behavioral and cognitive responses which may be maintaining the problem;
  4. adopt a healthy sleep routine which can promote healthy living.
  Hand-outs will be available for GPs to give to patients, but the structure of the intervention allows for treatment to be formulation-based so that particular issues raised in the consultation that might be maintaining symptom severity (e.g. avoidance) can be addressed.
  Arms: Integrated GP Care

SUMMARY:
PRINCE primary is cluster randomised waiting list controlled trial to evaluate the feasibility of an integrated approach to care in general practice for adults with persistent physical symptoms (PPS). PPS is defined as physical symptoms with no obvious underlying organic. 240 patients with PPS recruited from 8-12 GP practices in London will be randomised to the integrated care approach plus treatment as usual (TAU) or TAU alone. The integrated GP approach consists of providing GPs with a short cognitive behaviour therapy (CBT) skills training, ongoing supervision, as well as written and audio-visual materials/guidelines. In addition, participants randomised to the intervention group will receive tailored CBT-based self-help materials (i.e. written and audio-visual materials).

DETAILED DESCRIPTION:
Patients with PPS are often severely functionally impaired and. They consume large amounts of healthcare and welfare benefits. There is an accumulating body of evidence showing that cognitive behavioural interventions can reduce levels of symptoms and improve overall functioning in patients with PPS. CBT has demonstrated both short-term and long-term efficacy with small to medium effect sizes for PPS. Larger treatment effects have been reported for specific PPS syndromes, including non-cardiac chest pain, Irritable Bowel Syndrome (IBS), and Chronic Fatigue Syndrome (CFS).

General practitioners (GPs) play a major role in identifying and managing patients with PPS. A previous randomised parallel group pilot trial investigated the feasibility (i.e. recruitment, retention and acceptability) of implementing a primary care Symptoms Clinic for patients with PPS). The Symptoms Clinic comprised a structured set of consultations delivered by a specially trained GP with a strong interest in PPS. The intervention included exploring potential biological mechanisms underlying the PPS condition, empathetic support, and training patients in symptom-management (i.e. medication or cognitive behavioural techniques). The results indicated that the Symptoms Clinic was acceptable to the majority of patients randomised to the intervention group, and may have the potential to generate clinically significant benefits. However, this pilot study did not assess feasibility parameters referring to GPs' willingness to participate in the study and undergo specialised psychological training. Moreover, the intervention was carried out by only one GP, raising questions about the generalizability of the study.

Managing patients with PPS can be highly challenging in general practice. Although GPs recognise the treatment of PPS as a responsibility of primary care, previous studies show that GPs often feel powerless, frustrated and helpless when encountering these patients. Furthermore, GPs frequently report that factors such as time constraints and the lack of psychological training prevents them from effectively addressing patients' psychosocial needs and developing appropriate doctor-patient communication skills.

The aim of this study is to assess whether it is feasible to conduct an adequately powered future trial to evaluate the efficacy and cost-effectiveness of a CBT-based integrated GP care approach for treating patients with PPS (please refer to arms and interventions for more details).

ELIGIBILITY:
Patients that fit the eligibility criteria will be invited to take part in the study. Patients will be considered eligible for inclusion in this study if they fulfil all of the following criteria:

(i) have a PPS diagnosis (which are medically unexplained) (ii) are greater than or equal to 18 and less than or equal to 65 years old (iii) are registered with a GP practice in South London that has consented to taking part in PRINCE Primary (iv) have had 6 or more consultations in the last year (not necessarily for the same symptom or directly related to PPS (v) have given written informed consent, provided baseline data before randomisation and can speak and read English at a level adequate for participation in the.

Patients will be excluded from the study if the patient has:

(i) active psychosis (ii) drug or alcohol addiction as indicated in the patient's medical notes (iii) current benzodiazepine use exceeding the equivalent of 10mg diazepam per day (iv) had any psychotherapy treatment within the last year (not inclusive of general visits from community psychiatric teams) (v) dissociative seizures (vi) if they are at imminent risk of self-harm, after psychiatric/ psychological assessment (vii) taking part in the PRINCE Secondary study or the ACTIB Study (Everitt et al., 2015).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2015-05; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Feasibility: Willingness of clinicians to participate in the study (proportion of GPs that register within the study out of the GPs that are registered with the eligible practice) | 24 weeks post randomization
  The following definition of a feasibility study has been agreed by the Efficacy and Mechanism Evaluation (EME), Public Health Research (PHR), Health Technology Assessment (HTA) and Research for Patient Benefit (RfPB) programme: "Feasibility Studies are pieces of research done before a main study in order to answer the question "Can this study be done?". They are used to estimate important parameters that are needed to design the main study".
Feasibility: Willingness of patients to use the provided material given in 'integrated GP care' (self-help material). | 24 weeks post randomization
  The following definition of a feasibility study has been agreed by the Efficacy and Mechanism Evaluation (EME), Public Health Research (PHR), Health Technology Assessment (HTA) and Research for Patient Benefit (RfPB) programme: "Feasibility Studies are pieces of research done before a main study in order to answer the question "Can this study be done?". They are used to estimate important parameters that are needed to design the main study".
Feasibility: Willingness of practices and participants to be contacted about the study (Number (No.) of reply slips sent via the post to ask if the practice/participants would like to participate further information v No. of reply slips received back) | 24 weeks post randomization
  The following definition of a feasibility study has been agreed by the Efficacy and Mechanism Evaluation (EME), Public Health Research (PHR), Health Technology Assessment (HTA) and Research for Patient Benefit (RfPB) programme: "Feasibility Studies are pieces of research done before a main study in order to answer the question "Can this study be done?". They are used to estimate important parameters that are needed to design the main study".
Feasibility: Willingness of practices to be randomised (No. of eligible GP practices agreed consent v No. of GP practices not agreed to consent) | 24 weeks post randomization
  The following definition of a feasibility study has been agreed by the Efficacy and Mechanism Evaluation (EME), Public Health Research (PHR), Health Technology Assessment (HTA) and Research for Patient Benefit (RfPB) programme: "Feasibility Studies are pieces of research done before a main study in order to answer the question "Can this study be done?". They are used to estimate important parameters that are needed to design the main study".
Feasibility: Willingness of GP practices to be consent and be randomized as assessed by No. of eligible GP practices agreed consent v No. of GP practices not agreed to consent | 24 weeks post randomization
  The following definition of a feasibility study has been agreed by the Efficacy and Mechanism Evaluation (EME), Public Health Research (PHR), Health Technology Assessment (HTA) and Research for Patient Benefit (RfPB) programme: "Feasibility Studies are pieces of research done before a main study in order to answer the question "Can this study be done?". They are used to estimate important parameters that are needed to design the main study".
Feasibility: Follow-up rates and response rates to questionnaires (Sent questionnaires v completed questionnaires received at 12 and 24 weeks). | 24 weeks post randomization
  The following definition of a feasibility study has been agreed by the Efficacy and Mechanism Evaluation (EME), Public Health Research (PHR), Health Technology Assessment (HTA) and Research for Patient Benefit (RfPB) programme: "Feasibility Studies are pieces of research done before a main study in order to answer the question "Can this study be done?". They are used to estimate important parameters that are needed to design the main study".
Feasibility: Rate of eligible trial participants (Consort). The number of patients per practice that are initially screened for eligibility and the number per practice meeting the inclusion and exclusion criteria. | 24 weeks post randomization
  The following definition of a feasibility study has been agreed by the Efficacy and Mechanism Evaluation (EME), Public Health Research (PHR), Health Technology Assessment (HTA) and Research for Patient Benefit (RfPB) programme: "Feasibility Studies are pieces of research done before a main study in order to answer the question "Can this study be done?". They are used to estimate important parameters that are needed to design the main study".
Feasibility: Availability of data required and the usefulness and limitations of GP databases assessed qualitatively | 24 weeks post randomization
  The following definition of a feasibility study has been agreed by the Efficacy and Mechanism Evaluation (EME), Public Health Research (PHR), Health Technology Assessment (HTA) and Research for Patient Benefit (RfPB) programme: "Feasibility Studies are pieces of research done before a main study in order to answer the question "Can this study be done?". They are used to estimate important parameters that are needed to design the main study".
Feasibility: Willingness of participants to be consented and randomised (No. of positive reply slips received V No. of patients agreed to be screened, No. of eligible patients agreed consent v No. of eligible patients not agreed to consent) | 24 weeks post randomization
  The following definition of a feasibility study has been agreed by the Efficacy and Mechanism Evaluation (EME), Public Health Research (PHR), Health Technology Assessment (HTA) and Research for Patient Benefit (RfPB) programme: "Feasibility Studies are pieces of research done before a main study in order to answer the question "Can this study be done?". They are used to estimate important parameters that are needed to design the main study".

OTHER OUTCOMES:
Work and Social Adjustment Scale (WSAS) | 24 weeks post randomization
  a five-item scale with a range of scores from 0 to 40 (a higher score indicates more severe impairment) that is used to measure patients' own perceptions of the impact of PPS on their functioning in terms of work, home management, social leisure and private leisure activities, family and other relationships.
Patient Health Questionnaire-15 (PHQ-15) | 24 weeks post randomization
  a 15-item scale measuring somatic symptoms and taking values from 0 to 30.
Patient Health Questionnaire-9 (PHQ-9) | 24 weeks post randomization
  a 9-item scale measuring depressive symptoms taking values from 0 to 27, with scores of scores of 5, 10, 15, and 20 representing mild, moderate, moderately severe, and severe depression respectively (Kroenke, Spitzer & Williams, 2001).
Clinical Global Impression (CGI) | 24 weeks post randomization
  a nine-point scale measuring patient's perceived improvement, where 1 is completely recovered and 9 is could not get any worse
Satisfaction (Measure patients' self-rated satisfaction of the intervention) | 24 weeks post randomization
  Measure patients' self-rated satisfaction of the intervention.
Client Service Receipt Inventory (Measures health care service receipt, direct and indirect costs of illness, and cost effectiveness of intervention) | 24 weeks post randomization
  questionnaire detailing patient's use of services, including:
  * Use of care providers (yes/no and type)
  * Attendance at accident and emergency (yes/no)
  * Use of diagnostic tests (yes/no and type)
  * Working hours, occupation and days absent from work
  * Receipt of benefits (yes/no and type)
GPs knowledge Questionnaire | 24 weeks post randomization
  Measures GP knowledge: 10 true of false statements testing the GP's knowledge of PPS (maximum score of 11)
GP's Confidence Questionnaire | 24 weeks post randomization
  Measures GP confidence: and a ten-item scale testing their confidence treating PPS (minimum score 10 and maximum score 70)
Cognitive Behavioural Responses Questionnaire (CBRQ) | 24 weeks post randomization
  measure of putative mediators of cognitive change including:
  * fear avoidance (range 0-24),
  * catastrophizing (range 0-16),
  * damage avoidance (range 0-20),
  * embarrassment avoidance (range 0-24),
  * symptom focusing (range 0-24),
  * all or nothing behaviour (range 0-20) and avoidance behaviour (range 0-32) (Reme, Stahl & Chalder, 2011)
EuroQol - 5 Dimensions - 5 Levels (EuroQol-5D-5L) | 24 weeks post randomization
  a 5-item scale measuring health, taking from 5 to 25. Additionally, patients rate their own perceptions of their current health on a scale of 0 to 100 (Brooks, 1996).

CONTACTS AND LOCATIONS:
Overall Officials: Trudie Chader, PhD, Principal Investigator — King's College London
Locations (1):
- Kings College London, London, United Kingdom

REFERENCES:
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-15: validity of a new measure for evaluating the severity of somatic symptoms. Psychosom Med. 2002 Mar-Apr;64(2):258-66. doi: 10.1097/00006842-200203000-00008. PMID 11914441
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] Brooks R. EuroQol: the current state of play. Health Policy. 1996 Jul;37(1):53-72. doi: 10.1016/0168-8510(96)00822-6. PMID 10158943
- [Background] Kleinstauber M, Witthoft M, Hiller W. Efficacy of short-term psychotherapy for multiple medically unexplained physical symptoms: a meta-analysis. Clin Psychol Rev. 2011 Feb;31(1):146-60. doi: 10.1016/j.cpr.2010.09.001. Epub 2010 Sep 16. PMID 20920834
- [Background] Nimnuan C, Hotopf M, Wessely S. Medically unexplained symptoms: an epidemiological study in seven specialities. J Psychosom Res. 2001 Jul;51(1):361-7. doi: 10.1016/s0022-3999(01)00223-9. PMID 11448704
- [Background] Sharpe M, Stone J, Hibberd C, Warlow C, Duncan R, Coleman R, Roberts R, Cull R, Pelosi A, Cavanagh J, Matthews K, Goldbeck R, Smyth R, Walker A, Walker J, MacMahon A, Murray G, Carson A. Neurology out-patients with symptoms unexplained by disease: illness beliefs and financial benefits predict 1-year outcome. Psychol Med. 2010 Apr;40(4):689-98. doi: 10.1017/S0033291709990717. Epub 2009 Jul 23. PMID 19627646
- [Background] Altayar O, Sharma V, Prokop LJ, Sood A, Murad MH. Psychological therapies in patients with irritable bowel syndrome: a systematic review and meta-analysis of randomized controlled trials. Gastroenterol Res Pract. 2015;2015:549308. doi: 10.1155/2015/549308. Epub 2015 Jan 31. PMID 25802514
- [Background] Burton C, Weller D, Marsden W, Worth A, Sharpe M. A primary care Symptoms Clinic for patients with medically unexplained symptoms: pilot randomised trial. BMJ Open. 2012 Feb 9;2(1):e000513. doi: 10.1136/bmjopen-2011-000513. Print 2012. PMID 22327629
- [Background] Johansen ML, Risor MB. What is the problem with medically unexplained symptoms for GPs? A meta-synthesis of qualitative studies. Patient Educ Couns. 2017 Apr;100(4):647-654. doi: 10.1016/j.pec.2016.11.015. Epub 2016 Nov 21. PMID 27894609
- [Background] Jonsbu E, Dammen T, Morken G, Moum T, Martinsen EW. Short-term cognitive behavioral therapy for non-cardiac chest pain and benign palpitations: a randomized controlled trial. J Psychosom Res. 2011 Feb;70(2):117-23. doi: 10.1016/j.jpsychores.2010.09.013. Epub 2010 Dec 3. PMID 21262413
- [Background] Kennedy TM, Chalder T, McCrone P, Darnley S, Knapp M, Jones RH, Wessely S. Cognitive behavioural therapy in addition to antispasmodic therapy for irritable bowel syndrome in primary care: randomised controlled trial. Health Technol Assess. 2006 Jun;10(19):iii-iv, ix-x, 1-67. doi: 10.3310/hta10190. PMID 16729918
- [Background] Kisely SR, Campbell LA, Skerritt P, Yelland MJ. Psychological interventions for symptomatic management of non-specific chest pain in patients with normal coronary anatomy. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD004101. doi: 10.1002/14651858.CD004101.pub3. PMID 20091559
- [Background] Moss-Morris R, Chalder T. Illness perceptions and levels of disability in patients with chronic fatigue syndrome and rheumatoid arthritis. J Psychosom Res. 2003 Oct;55(4):305-8. doi: 10.1016/s0022-3999(03)00013-8. PMID 14507540
- [Background] Salmon P, Peters S, Clifford R, Iredale W, Gask L, Rogers A, Dowrick C, Hughes J, Morriss R. Why do general practitioners decline training to improve management of medically unexplained symptoms? J Gen Intern Med. 2007 May;22(5):565-71. doi: 10.1007/s11606-006-0094-z. PMID 17443362
- [Background] van Dessel N, den Boeft M, van der Wouden JC, Kleinstauber M, Leone SS, Terluin B, Numans ME, van der Horst HE, van Marwijk H. Non-pharmacological interventions for somatoform disorders and medically unexplained physical symptoms (MUPS) in adults. Cochrane Database Syst Rev. 2014 Nov 1;2014(11):CD011142. doi: 10.1002/14651858.CD011142.pub2. PMID 25362239
- [Background] White PD, Goldsmith KA, Johnson AL, Potts L, Walwyn R, DeCesare JC, Baber HL, Burgess M, Clark LV, Cox DL, Bavinton J, Angus BJ, Murphy G, Murphy M, O'Dowd H, Wilks D, McCrone P, Chalder T, Sharpe M; PACE trial management group. Comparison of adaptive pacing therapy, cognitive behaviour therapy, graded exercise therapy, and specialist medical care for chronic fatigue syndrome (PACE): a randomised trial. Lancet. 2011 Mar 5;377(9768):823-36. doi: 10.1016/S0140-6736(11)60096-2. Epub 2011 Feb 18. PMID 21334061
- [Background] Bermingham SL, Cohen A, Hague J, Parsonage M. The cost of somatisation among the working-age population in England for the year 2008-2009. Ment Health Fam Med. 2010 Jun;7(2):71-84. PMID 22477925
- [Background] Everitt H, Landau S, Little P, Bishop FL, McCrone P, O'Reilly G, Coleman N, Logan R, Chalder T, Moss-Morris R; ACTIB trial team. Assessing Cognitive behavioural Therapy in Irritable Bowel (ACTIB): protocol for a randomised controlled trial of clinical-effectiveness and cost-effectiveness of therapist delivered cognitive behavioural therapy and web-based self-management in irritable bowel syndrome in adults. BMJ Open. 2015 Jul 15;5(7):e008622. doi: 10.1136/bmjopen-2015-008622. PMID 26179651
- [Background] Chalder T, Wallace P, Wessely S. Self-help treatment of chronic fatigue in the community: A randomized controlled trial. British Journal of Health Psychology 1997;2(3):189-97. doi: https://doi.org/10.1111/j.2044-8287.1997.tb00535.x
- [Background] Reme SE, Stahl D, Kennedy T, Jones R, Darnley S, Chalder T. Mediators of change in cognitive behaviour therapy and mebeverine for irritable bowel syndrome. Psychol Med. 2011 Dec;41(12):2669-79. doi: 10.1017/S0033291711000328. Epub 2011 Apr 11. PMID 21477419
- [Derived] Patel M, James K, Moss-Morris R, Ashworth M, Husain M, Hotopf M, David AS, McCrone P, Landau S, Chalder T; PRINCE Primary trial team. BMC family practice integrated GP care for patients with persistent physical symptoms: feasibility cluster randomised trial. BMC Fam Pract. 2020 Oct 7;21(1):207. doi: 10.1186/s12875-020-01269-9. PMID 33028243
- [Derived] Patel M, James K, Moss-Morris R, Husain M, Ashworth M, Frank P, Ferreira N, Mosweu I, McCrone P, Hotopf M, David A, Landau S, Chalder T. Persistent physical symptoms reduction intervention: a system change and evaluation (PRINCE)-integrated GP care for persistent physical symptoms: protocol for a feasibility and cluster randomised waiting list, controlled trial. BMJ Open. 2019 Jul 23;9(7):e025513. doi: 10.1136/bmjopen-2018-025513. PMID 31340956